CLINICAL TRIAL: NCT06282926
Title: Role of Three-dimensional Echocardiography Knowledge-based Reconstruction in Monitoring Right Ventricle Remodelling Following Tetralogy of Fallot Repair
Brief Title: Role of 3D Echocardiography Knowledge-based Reconstruction in ACHD
Status: Active, not recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 324811
Record Dates: First submitted 2023-08-10; First posted 2024-02-28 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group 1: Healthy adult volunteers
  Interventions: Diagnostic Test: Echocardiography assessment
- Group 2: ACHD patients with repaired Tetralogy of Fallot and known moderate or severe pulmonary regurgitation
  Interventions: Diagnostic Test: Echocardiography assessment

INTERVENTIONS:
Diagnostic Test: Echocardiography assessment — Group 1 will have healthy adult volunteers recruited at the workplace following specific criteria to participate in the study. A research cardiac ultrasound protocol to assess the RV will be performed at two different visits, with a maximum interval of two weeks between them.
  Group 2 will have ACHD patients with known moderate or severe pulmonary regurgitation after ToF repair, following specific criteria to participate in the study. This group of patients will be studied in two separate visits. The patients will be recruited during the first visit when attending to an existing hospital appointment for ACHD CMR. A research cardiac ultrasound protocol to assess the RV will be performed on the same day, either before or after the CMR. For all patients who will have a second follow-up visit at the ACHD outpatient clinic within a maximum interval of one year, the same research protocol will be performed, in addition to the usual cardiac ultrasound.
  Other Names: Cardiac Magnetic Resonance

SUMMARY:
The main objective of this study is to evaluate the reproducibility and accuracy of TTE-3DKBR in assessing RV volume and EF compared to the reference method of CMR in a group of ACHD patients with known moderate or severe PR after ToF repair.

As part of the validation study, the reproducibility of the TTE-3DKBR in assessing RV volume and EF will also be tested in a group of healthy adult volunteers. Additionally, TTE-3DKBR evaluation will be compared in both groups to the conventional 2D echocardiography measurements used in routine clinical practice, such as tricuspid annular plane systolic excursion (TAPSE), tissue Doppler imaging (TDI), fractional area change (FAC), and global longitudinal strain (GLS).

Another objective of the study is also to evaluate the effects of chronic RV volume overload with an interval of one-year follow-up using TTE-3DKBR and compare it with the conventional non-geometric echocardiography measurements, particularly with GLS.

The study will end when the required number of patients have been enrolled and when the last subject undergoes the research dataset acquisition. The study may be terminated prematurely if it becomes apparent that the recruitment target cannot be met within the projected recruitment phase.

DETAILED DESCRIPTION:
Tetralogy of Fallot (ToF) is a complex pathophysiology characterised by different factors that affect the right ventricle (RV) performance. Before surgical repair in childhood, the RV is exposed to pressure load with associated abnormal RV outflow tract (RVOT) hypertrophy and myocardial damage related to prolonged cyanosis. After surgical repair involving a pulmonary valve (PV) transannular patch, the RV may experience chronic volume overload due to significant pulmonary regurgitation (PR). The effects of chronic volume overload often found in adult congenital heart disease (ACHD) patients frequently result in progressive RV dilatation with abnormal geometry and RV dysfunction with associated electromechanical dyssynchrony. All this often leads to re-intervention with PV replacement. In asymptomatic patients with severe PR, the 2020 European ACHD guidelines recommendation for PV replacement gives a class 2a recommendation and evidence level C in cases of progressive RV systolic dysfunction and/or dilatation with a RV indexed end-diastolic volume (EDVi) ≥160 mL/m2, and/or a RV indexed end-systolic volume (ESVi) ≥80 mL/m2. The guidelines also mentioned gaps regarding the need for more longitudinal imaging data to optimise time for re-intervention because the possibility for RV remodelling is, at some point, irreversible.

CMR is widely recognised in the literature as the reference standard imaging technique for accurately quantifying RV volume and ejection fraction (EF) in the ACHD population. However, unlike transthoracic echocardiography (TTE), CMR is not the first-line test used in daily clinical practice.

The echocardiographic requirement of conventional multiple non-geometric (tricuspid annular plane systolic excursion, tissue Doppler imaging, global longitudinal strain) and geometric two-dimensional (2D) parameters (fractional area change, three-dimensional volume and EF) for a more accurate RV size and systolic function assessment is consensual in the literature with global longitudinal strain (GLS) emerging as a simple and effective tool for the management of repaired ToF patients. Also, it is known that conventional three-dimensional (3D) echocardiography systematically underestimates RV volumes and overestimates EF. Therefore, CMR and conventional 3D echo should not be used interchangeably.

Alternatively, 3D knowledge-based reconstruction derived from 2D echocardiography (TTE-3DKBR) has shown to be a valuable tool for RV volume and EF assessment that can complement CMR and maximise the available resources in clinical practice. The literature on TTE-3DKBR in children and adults with ToF indicates a high correlation with CMR, and its potential for clinical follow-up in repaired ToF patients may be relevant. However, the recommendations of the expert consensus documents are also clear that further validation studies are needed before its implementation in clinical practice.

The current longitudinal study aims to further the role of TTE-3DKBR in evaluating the effects of chronic RV volume overload in ACHD repaired ToF patients by assessing its reproducibility and accuracy against CMR and conventional echocardiography measurements, particularly with standard GLS.

ELIGIBILITY:
Inclusion Criteria:

Group 1 of healthy adult volunteers - Minimum aged of 18 years old without evidence of structural heart disease.

Group 2 of ACHD patients - ACHD patient minimum aged of 18 years old with diagnosis of moderate or severe pulmonary regurgitation after ToF repair.

Exclusion Criteria:

Group 1 of healthy adult volunteers - No informed consent, evidence of structural heart disease.

Group 2 of ACHD patients - No informed consent, pacemaker or defibrillator non-compatible with CMR, limited echocardiographic images for image acquisition, and evidence of moderate or severe right ventricle inflow and/or right ventricle outflow tract obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 of healthy adult volunteers
  Group 2 of ACHD patients with repaired Tetralogy of Fallot and known moderate or severe pulmonary regurgitation
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Evaluate the reproducibility and accuracy of TTE-3DKBR in assessing RV volume and EF compared to the reference method of CMR in a group of ACHD patients with known moderate or severe PR after ToF repair. | First year of the study
  To study what is the maximum considered acceptable mean difference between RV volumes measures between CMR and TTE-3DKBR.
Evaluate the effects of chronic RV volume overload in this population within one-year follow-up using TTE-3DKBR and compare it with the conventional non-geometric echocardiography measurement of GLS. | Second year of the study
  To study the predictive value of RV volumes using TTE-3DKBR to assess RV systolic dysfunction defined by GLS below -18%.

SECONDARY OUTCOMES:
Compare TTE-3DKBR evaluation to the conventional 2D echocardiography measurements used in routine clinical practice (TAPSE, TDI, FAC, and GLS). | First year of the study
  To study whether TTE-3DKBR values correlate with conventional 2D echocardiography measurements used in routine clinical practice (TAPSE, TDI, FAC and GLS).

CONTACTS AND LOCATIONS:
Overall Officials: Dario Luis Leal de Freitas, BSc, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided